CLINICAL TRIAL: NCT06085781
Title: HN-BIO: A Study of Head and Neck MRI and Tumor Microenvironment Biomarkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-BIO
Record Dates: First submitted 2023-10-09; First posted 2023-10-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pimonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Other): Participants who are to receive standard of care radiotherapy will have one biopsy and MRI scan before starting radiotherapy and during week two of radiotherapy. Participants will also have an the option to consent to an additional biopsy and MRI scan during week 4 of radiotherapy. Oral pimonidazole will be taken the night before each biopsy.
  Interventions: Other: fMRI; Other: Oral Pimonidazole
- Cohort B (Other): Participants who are to receive standard of care curative surgery will have an MRI scan within one week prior to surgery. Tumor tissue from the surgery will also be collected for research. Oral pimonidazole will be taken the night before surgery.
  Interventions: Other: fMRI; Other: Oral Pimonidazole

INTERVENTIONS:
Other: fMRI — Functional Magnetic Resonance Imaging
Other: Oral Pimonidazole — 200 mg and 300 mg tablets

SUMMARY:
The purpose of this study is to explore biomarker development in patients with newly diagnosed Head and neck squamous cell carcinoma (HNSCC) receiving curative therapy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be assigned to Cohort A or Cohort B.

Cohort A will recruit up to 40 patients planned to receive curative radiotherapy for HNSCC. Patients will undergo a baseline fMRI (Functional Magnetic Resonance Imaging) scan and within 72 hours a biopsy of the primary tumor will be performed in out-patient clinic. In week 2 of radiotherapy a further biopsy of the primary site will be performed with a paired fMRI performed within 72 hours prior to biopsy assess evolving changes in imaging and tumor microenvironment biomarkers during radiotherapy. A further optional biopsy and paired MRI scan in week 4 will be considered for patients who are tolerating therapy without toxicities. 16-24 hours prior to each biopsy the volunteer will take oral pimonidazole.

Cohort B will recruit up to 20 patients planned to receive curative surgery for HNSCC. Each patient will undergo a baseline fMRI scan performed within one week prior to surgery. At time of initial consent they will receive a prescription for oral pimonidazole hydrochloride which they will be asked to take the 16-24 hours before planned surgery. Following surgery whole tumor samples will be processed to permit spatial reconstruction of pimonidazole staining hypoxia to correlate with fMRI imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Histologically proven Head and Neck Squamous Cell carcinoma
* Primary or nodal disease > 3cm for biomarker imaging
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Planned for curative surgery or (chemo)radiotherapy
* Willingness to undergo repeat MRI imaging
* Able to receive and understand verbal and written information regarding study and able to give written informed consent
* Adequate renal function: Calculated creatinine clearance >/= 30ml/min
* Be able to lie comfortably on back for 1 hour

Exclusion Criteria:

* As judged by investigator evidence of systemic disease that makes unsuitable for study
* Contra-indication for serial MRI scans
* Previous solid tumor treated within last 5 years
* Pregnancy
* History of gadolinium contrast allergy
* Non-reversible clotting abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in tumor microenvironment during radiotherapy | Prior to radiotherapy, week 2 and week 4 of radiotherapy
  Repeat biopsy will be analyzed for haematoxylin and eosin (H&E), pimonidazole (monoclonal IgG1 antibody, Hypoxyprobe MAb1), endogenous proteins associated with hypoxia and/or immune infiltrate, DNA, and RNA.
Change in fMRI during radiotherapy | Prior to radiotherapy, week 2 and week 4 of radiotherapy
  Assessed through hypoxic regions visible on imaging scans

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada